CLINICAL TRIAL: NCT03188107
Title: Interrater and Intrarater Reliability of Infant Motor Profile: Assessing Motor Profiles of Risky Infants
Brief Title: Interrater Reliability of Infant Motor Profile
Acronym: IMP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayse Numanoglu Akbas, Pt, PhD, Abant Izzet Baysal University
Other Study IDs: AbantIbu01
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Premature Infants; Cerebral Palsy; Down Syndrome; Metabolic Disorders; Spina Bifida; Low; Birthweight, Extremely (999 Grams or Less)
Keywords: Risky Infant; Cerebral Palsy; Down Syndrome; Spina Bifida; Infant Motor Profile
MeSH Terms: conditions — Premature Birth; Cerebral Palsy; Down Syndrome; Metabolic Diseases; Spinal Dysraphism; Birth Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Risky Infants: Infants that have risk of developing motor impairment, or infants diagnosed as Spina Bifida, Down Syndrome ect.
  Interventions: Other: Video based assessment
- Healthy Infants: Healthy infants that have normal motor development
  Interventions: Other: Video based assessment

INTERVENTIONS:
Other: Video based assessment — All the infants included in this study will be assessed with Infant Motor Profile based on video recording.

SUMMARY:
The aim of this study is to assess risky infants (or diagnosed infants) with Infant Motor Profile, and analyze interrater and intrarater reliability of this test.

DETAILED DESCRIPTION:
It is very hard to assess risky infants because of many problems like lack of cooperation, crying, discomfort ect. But with "Infant Motor Profile (IMP)" it is possible to assess motor behavior of risky infants in their daily environment. The assessment relays on video recordings so after recording the motor behavior many people can score the same children many times to have a certain idea about the infant. With this tool it could be easier to set a therapy program after determining the basic motor problem. In Turkey there are a lot of risky infants which later have diagnosed with Cerebral Palsy, Metabolic Disorders and other diseases. Also there are a lot of infants with Down Syndrome (DS) and Spina Bifida (SB). It has been known motor development is impaired with different childhood conditions but there is less information in literature about motor development of children with SB, DS and other diseases. With this study motor status of risky infants between 3- 24 months old will be explored, interrater and intrarater reliability of Infant Motor Profile will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Cerebral Palsy
* Clinical Diagnosis of Down Syndrome
* Clinical Diagnosis of Spina Bifida

Exclusion Criteria:

* Uncontrolled Epilepsy
* Severe Congenital Disorders

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study population consists of risky infants (premature infants, low birth weighted infants, infants with spina bifida or down syndrome
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Infant Motor Profile | Infants will be assessed at baseline and 3 months later from the first assessment.
  Video recording based assessment of motor status

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe NUMANOĞLU AKBAŞ, PhD, Principal Investigator — Abant Izzet Baysal University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Heineman KR, Bos AF, Hadders-Algra M. Infant Motor Profile and cerebral palsy: promising associations. Dev Med Child Neurol. 2011 Sep;53 Suppl 4:40-5. doi: 10.1111/j.1469-8749.2011.04063.x. PMID 21950393